CLINICAL TRIAL: NCT01231802
Title: A Comparative, Multicenter, Open-Label, Randomized, Phase 2 Study of the Safety and Antitumor Activity of Oral Eniluracil + 5 Fluorouracil + Leucovorin Versus Capecitabine Monotherapy in Subjects With Metastatic Breast Cancer
Brief Title: Study of Eniluracil + 5-Fluorouracil (5-FU) + Leucovorin Versus Capecitabine in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adherex Technologies, Inc. (Industry)
Responsible Party: Gray Kirby/Clinical Project Manager, Adherex Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHX-03-202
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eniluracil; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Eniluracil/5-FU/Leucovorin (Experimental): Arm 1: (weekly, 28-day cycle): Approximately eighty subjects will orally self-administer eniluracil approximately 13 hr (range of 11-16 hr) before receiving 5 FU and leucovorin. The next day they will orally self-administer 5-FU and leucovorin. On the third day, they will orally self-administer leucovorin. The regimen is taken once per week for three consecutive weeks followed by one-week off-treatment.
  Interventions: Drug: Eniluracil; Drug: 5-Fluorouracil; Drug: Leucovorin
- Arm 2: Capecitabine (Active Comparator): Arm 2: (bid daily, 21-day cycle): Approximately sixty subjects will self-administer oral capecitabine (1000 mg/m2) twice daily (12 hr apart) for 14 consecutive days followed by 7 days off-treatment
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Eniluracil — Eniluracil (40 mg) orally at 18:00 ± 1 hour (6:00 PM) on Days 1, 8, & 15
  Arms: Arm 1: Eniluracil/5-FU/Leucovorin
Drug: 5-Fluorouracil — 5-FU (30 mg/m2) orally at 7:00 AM ± 1 hour on Days 2, 9, & 16
  Arms: Arm 1: Eniluracil/5-FU/Leucovorin
Drug: Leucovorin — Leucovorin (30 mg) orally at 7:00 AM ± 2 hours on Days 2, 3, 9, 10, 16, & 17
  Arms: Arm 1: Eniluracil/5-FU/Leucovorin
Drug: Capecitabine — Capecitabine (1000 mg/m2) twice daily (12 hr apart) for 14 consecutive days followed by 7 days off-treatment
  Arms: Arm 2: Capecitabine

SUMMARY:
The purpose of the study is to determine if eniluracil/5-FU/leucovorin in metastatic breast cancer (MBC) may have efficacy and tolerability advantages over capecitabine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic (Stage IV) adenocarcinoma of the breast
* Prior exposure to anthracyclines either in the neoadjuvant/adjuvant setting, or as treatment for metastatic disease
* Either evidence of a recurrence or development of metastatic disease at least 12 months after the last dose of a taxane as neoadjuvant/adjuvant therapy, or evidence of disease progression while receiving a taxane for metastatic disease
* ECOG Performance Status of 0 or 1
* Measurable disease according to RECIST 1.1 Criteria
* Adequate renal, hematologic, and hepatic function
* Negative pregnancy test and willing to use effective contraception
* Willing to avoid any other dose or form (iv, oral, or topical) of 5 FU or related derivatives for 8 weeks following the last dose of eniluracil
* Willing to be closely monitored for changes in coagulation parameters (prothrombin time and/or international normalized ratio [INR] values) if receiving concomitant warfarin

Exclusion Criteria:

* Pregnant or lactating females
* Prior treatment with capecitabine
* More than one prior chemotherapy regimen for metastatic disease
* Prior radiation must not have included ≥ 30% of major bone marrow-containing areas (pelvis, lumbar spine). If prior radiation was < 30%, then a minimum interval of 6 weeks must be allowed between the last radiation treatment and administration of either study arm.
* Currently receiving anti-cancer therapy
* Residual ≥ Grade 2 clinically significant side effects (excluding alopecia) associated with prior radiotherapy, chemotherapy, and investigational treatments
* Unstable CNS metastases. However, subjects that are asymptomatic and off systemic steroids and anticonvulsants for at least 3 months are not excluded.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, ulcerative colitis, recent history of GI bleeding or perforation
* History of other malignancy, except subjects who have been disease-free for 5 years or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety
* Known history or clinical evidence of leptomeningeal carcinomatosis
* Active or uncontrolled infection
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Known history of uncontrolled or symptomatic angina, arrhythmia or congestive heart failure
* Concurrent treatment with an investigational agent
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication
* Taking phenytoin
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to capecitabine, fluorouracil, leucovorin, or any excipients
* Known dihydropyrimidine dehydrogenase (DPD) deficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-08 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 7.5 months

SECONDARY OUTCOMES:
To compare the tolerability and toxicity of orally administered eniluracil/5 FU/leucovorin regimen vs. capecitabine monotherapy | 7.5 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (2):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - The Methodist Hospital Cancer Center, Houston, Texas
- Russia (14):
  - Arkhangelsk Regional Clinical Oncology Center, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology, Chelyabinsk
  - Clinical Oncology Center #1, Krasnodar
  - Moscow Hertzen Oncology Research Institute, Moscow
  - Russian Oncological Research Center n.s. Blokhin, Moscow
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Pyatigorsk Oncology Center, Pyatigorsk
  - Republic Oncology Center, Republic of Karelia
  - City Clinical Oncology Center, Saint Petersburg
  - Laboratory of Thoracic Oncology of Research Institute of Pulmonary at St. Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - Leningrad Regional Oncology Center, Saint Petersburg
  - Road Clinical Hospital of the Russian Railways, Saint Petersburg
  - Oncology Center No. 2 Krasnodar Regional Healthcare Dept, Sochi
  - Stavropol Regional Clinical Oncology Center, Stavropol

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241